CLINICAL TRIAL: NCT06323226
Title: The Impact of Sepsis on Long-term Outcomes in Critical Ill Children With Sepsis
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Professor, West China Hospital
Other Study IDs: 2024-312-1
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Children, Only
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is conducted in critically ill children with sepsis with a five years follow-up. We aim to investigate the impact of sepsis on long-term outcomes including growth, neurodevelopment, survival rate, quality of life.

ELIGIBILITY:
Inclusion Criteria:

We included critically ill children with sepsis who successfully discharged from pediatric Intensive care units, age < 16 years.

We also included age, sex, illness severity matched critically ill children as control group.

Exclusion Criteria:

We excluded children with underlying diseases, cancer, hematologic malignancy.

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We included critically ill children with sepsis who successfully discharged from pediatric intensive care units and age < 16 years. Age, sex, and illness severity matched critically ill children would be included as control group.
  Children with underlying diseases, cancer, and hematologic malignancy would be excluded.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | Five years
  Rate of death in 5-years follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China